CLINICAL TRIAL: NCT07128459
Title: Lip Reduction Surgery for Port-wine Macrocheilia: a Retrospective Single-center Clinical Study
Brief Title: Lip Reduction Surgery for Port-wine Macrocheilia
Acronym: macrocheilia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Gang Ma, Associate Chief Physician, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SH9H-2025-T313-1
Record Dates: First submitted 2025-08-13; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Port Wine Stains
MeSH Terms: conditions — Hemangioma, Capillary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with port-wine macrocheilia who underwent lip reduction surgery using the five-step method (Experimental)
  Interventions: Procedure: The Five-Step lip reduction surgery

INTERVENTIONS:
Procedure: The Five-Step lip reduction surgery — The Five-Step lip reduction surgery: (1) measurement and design; (2) incision and reduction of lip volume; (3) fixation and shape of the dry lip; (4) fixation and shape of the skin (the SMISS approach); (5) shaping of the wet lip mucosa (the SMISS approach).

SUMMARY:
Patients with port-wine stains often develop macrocheilia, however, there is currently no effective treatment to significantly reduce the three-dimensional volume increase of the lips. This article presents a simplified "five-step" approach based on clinical experience, designed to assist inexperienced surgeons in performing this surgery effectively.

ELIGIBILITY:
Inclusion Criteria: 1. Patients with port-wine macrocheilia. 2. Patients that underwent lip reduction surgery. 3. Age at surgery: ≥3 years and ≤70 years.

Exclusion Criteria: 1. Patients without port-wine macrocheilia. 2. Missing/incomplete baseline patient information. 3. Patients without postoperative photographs.

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
the Visual Analog Scale | From enrollment to the end of treatment in 6 months to one year

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Ninth People's Hospital, Shanghai Jiao Tong University, School of Medicine, Shanghai, China